CLINICAL TRIAL: NCT07279038
Title: Symptom Evaluation and Quantification for Unified Outcomes and Individualized Assessment: Pivotal Clinical Validation Phase
Brief Title: Pivotal U.S. Clinical Validation of AI-COA® for Depression and Anxiety
Acronym: SEQUOIA-3
Status: Not yet recruiting | Type: Observational
Sponsor: Deliberate Solutions Inc. (Industry)
Collaborators: Baylor College of Medicine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: SEQUOIA-3
Record Dates: First submitted 2025-12-07; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Depression Disorders; Anxiety Disorders
Keywords: depression assessment; anxiety assessment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — audiovideo recordings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a large-scale pivotal clinical validation of the AI-COA® software device. The purpose is to confirm the tool's accuracy and performance across a demographically diverse population of adults with Major Depressive Disorder (MDD), ensuring it functions fairly and reliably across different subgroups.

DETAILED DESCRIPTION:
The SEQUOIA-3 study is a Comprehensive U.S. Clinical Validation of the AI-generated Clinical Outcome Assessment (AI-COA®) for depression and anxiety. This observational study supports the clinical validation of a digital tool intended to measure depression severity using audiovisual data from clinical interviews. The study builds on previous research to establish the tool's validity for regulatory qualification.

Key elements of the study include:

Diverse Enrollment: The study will prospectively enroll a large, stratified sample to ensure adequate representation across sex, race, and ethnicity, as well as a full range of symptom severity (from remission to severe).

Validation: The software's severity scores will be compared against a "ground truth" standard derived from the consensus of independent human raters.

Remote Assessment: Participants will complete standard clinical interviews and self-report measures via secure video conferencing.

The results will be used to demonstrate the tool's generalizability and its ability to provide unbiased assessments across different patient populations.

ELIGIBILITY:
Inclusion Criteria:

* English fluency
* 18 to 65 years of age.
* Diagnosed with MDD or MDE (Includes Remission, HAM-D <= 7)
* Starting, or has started, a new treatment for depression or anxiety within 2-3 weeks of enrollment
* Access to a laptop or other computer with a well functioning microphone and webcam, and a stable Internet connection
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Resides in the United States at the time of consent and during completion of study

Exclusion Criteria:

* Any cognitive impairment that limits ability to provide informed consent or authorization
* Vulnerable or protected populations (e.g. prisoners)
* Impairment that would prevent participants from completing an online survey and/or engaging in clinician assessment interviews (e.g., visual impairment, motor impairment, hearing impairment)
* Acute intoxication at the time of the assessments
* Concurrent medication/treatment:

  * Receiving any fast-acting treatment for depression or anxiety (e.g. ketamine, psychedelics, deep brain stimulation, etc.) in between initial baseline assessment (A1) and Restest (A2) , or in between Follow up assessment (B1) and Retest (B2)
  * Anxiolytics: Use of benzodiazepines or other anxiety-reducing medications that could affect speech or motor activity, within the past 4 weeks.
  * Antipsychotics and Mood Stabilizers: Medications that can alter cognitive and motor functions, within the past 6 weeks.
  * Stimulants: Use of medications like methylphenidate or amphetamines that affect energy levels and behavior, within the past 2 weeks
  * Epilepsy medication: seizure activity or medication side effects that may alter behavior, within the past 4 weeks.
* Any history or evidence of any of the following conditions:

  * Neurodevelopmental, Neurocognitive, Neurodegenerative or movement disorders including, but not limited to:
  * Tourette's syndrome
  * Multiple Sclerosis
  * Amyotrophic Lateral Sclerosis
  * Parkinson's Disease
  * Stroke
  * Traumatic Brain Injury
  * Facial paralysis.
* Conditions with vocal cord impact:

  * Vocal cord injury or cerebrovascular accident or head trauma with residual dysarthria in the past year
  * Disorders that may impact vocal cords such as acute or chronic laryngitis, vocal cord paresis or paralysis, or spasmodic dysphonia
  * Past or active heavy smokers (an average of >20 cigarettes per day)
* Schizophrenia Spectrum and Other Psychotic Disorders:

  * Individuals with a current or past diagnosis of Schizophrenia, Schizoaffective Disorder, or other psychotic disorders, including Delusional Disorder and Brief Psychotic Disorder.
  * Current hypomanic episode as defined by DSM-5 criteria. This includes those with Bipolar I Disorder, Bipolar II Disorder, or Cyclothymic Disorder who are not in a stable mood state at the time of assessment.
  * Chronic Pain Conditions: Such as fibromyalgia, which may affect facial expressions and vocal tone.
  * Prosthetic Facial Devices: Could affect facial recognition algorithms. Cosmetic Procedures: Such as Botox injections or facelifts that can impact facial expressions.
  * Dental Work: Major procedures that might affect speech.
* Participants who have previously participated in another research project by Deliberate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with MDD or MDE
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2027-03-01 (Estimated); Primary Completion 2029-08-28 (Estimated); Study Completion 2029-08-28 (Estimated)

PRIMARY OUTCOMES:
HAM-D ICC | Baseline
  Concordance of HAM-D score between model and human raters

SECONDARY OUTCOMES:
MADRS ICC | Baseline
  Concordance of MADRS score between model and human raters
HAM-A ICC | Baseline
  Concordance of HAM-A score between model and human raters

CONTACTS AND LOCATIONS:
Overall Officials: Marc Aafjes, Principal Investigator — Deliberate Solutions Inc.
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No